CLINICAL TRIAL: NCT03893630
Title: Role of Aspirin in Maternal Endothelial Dysfunction and Uterine Artery Blood Flow in Women at Risk for Preeclampsia
Brief Title: Role of ASpirin in Placental and Maternal Endothelial Cell Regulation IN Pre-eclampsia
Acronym: ASPERIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John O'Brien, MD (Other)
Responsible Party: Sponsor-Investigator, John O'Brien, MD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 47841
Record Dates: First submitted 2019-03-01; First posted 2019-03-28 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Pre-Eclampsia
Keywords: aspirin; pulsatility index; doppler; uterine; acetylsalicylic acid; preeclampsia; blood pressure
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control Group (Active Comparator): Patients will receive standard of care.
  Interventions: Other: Control
- Acetylsalicylic Acid 81mg (Experimental): Patients will receive low dose (81mg) acetylsalicylic acid (Aspirin).
  Interventions: Drug: Acetylsalicylic Acid 81 mg
- Acetylsalicylic Acid 162mg (Experimental): Patients will receive low dose (162mg) acetylsalicylic acid (Aspirin).
  Interventions: Drug: Acetylsalicylic Acid 162 mg

INTERVENTIONS:
Drug: Acetylsalicylic Acid 81 mg — Patients will receive 81mg acetylsalicylic acid daily, initiated between 11 and 16 weeks of gestation and continued until 36 weeks of gestation.
  Other Names: Aspirin
  Arms: Acetylsalicylic Acid 81mg
Drug: Acetylsalicylic Acid 162 mg — Patients will receive 162mg acetylsalicylic acid daily, initiated between 11 and 16 weeks of gestation and continued until 36 weeks of gestation.
  Other Names: Aspirin
  Arms: Acetylsalicylic Acid 162mg
Other: Control — Standard of Care
  Arms: Control Group

SUMMARY:
Endothelial dysfunction and defective placental vascularization are hypothesized to be significant causes of preeclampsia. In preeclampsia, due to vascular endothelial dysfunction, vasoconstriction and platelet activation can result in severe features which alter pregnancy outcomes. However, studies have shown that acetylsalicylic acid (Aspirin) can decrease endothelial dysfunction leading to decreased platelet aggregation which reduces adverse outcomes. The objective of our study is to determine if Aspirin has a dose-dependent response for modifying biomarkers reflective of maternal endothelial dysfunction when indicated for preeclampsia prevention in a cohort of women identified at risk for developing preeclampsia.

Pregnant women who are at risk for preeclampsia will be randomized to receive either 81mg Aspirin or 162mg Aspirin daily starting from 11-16 weeks of gestation until 36 weeks of gestation. A third, control group of women at low risk for preeclampsia will not receive aspirin. All women will be assessed with uterine artery Doppler studies and mean arterial blood pressures at three time points during pregnancy. Blood, urine, and cord blood samples will also be collected.

DETAILED DESCRIPTION:
Eligible women will be identified in the late first or early second trimesters. Once recruited, women will be randomly assigned to either 81 mg or 162 mg per day dosing schedules. The randomization scheme will vary based on the body mass index (BMI) with separate schemes for women <=30 kg/m2 versus >30 kg/m2. Ultrasonographic assessment of biophysical biomarkers will be obtained at 11-16 weeks, 18-22 weeks, and 28-32 weeks gestation. Biologic samples of serum and urine will be obtained at the 11-16 week and 28-32 week visit. Upon delivery, cord blood and a placental specimen will also be obtained. Medication treatment will continue until 36 weeks gestation. Pregnancy and neonatal outcome data will be recorded.

ELIGIBILITY:
Inclusion Criteria (control)

• No risk factors for preeclampsia

Inclusion Criteria (pre-eclampsia)

* History of preterm preeclampsia
* Chronic hypertension
* Type 1 and Type 2 diabetes
* Renal diseases
* Autoimmune disease

Exclusion Criteria

* Pregnant women younger than 18 years or older than 45 years
* Multiple gestations
* History of allergy (urticaria or anaphylaxis) to aspirin or aspirin-related products asthma that worsens after aspirin use
* Patients with gastrointestinal or genitourinary bleeding
* Patients with peptic ulcer disease
* Patients with severe liver dysfunction
* Patients who have undergone bypass surgery
* Patients on anticoagulant medication(s)
* Women with anomalous fetus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M O'Brien, MD, Principal Investigator — University of Kentucky; Katherine Vignes, MD, Study Chair — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Askie LM, Duley L, Henderson-Smart DJ, Stewart LA; PARIS Collaborative Group. Antiplatelet agents for prevention of pre-eclampsia: a meta-analysis of individual patient data. Lancet. 2007 May 26;369(9575):1791-1798. doi: 10.1016/S0140-6736(07)60712-0. PMID 17512048
- [Background] Roberge S, Bujold E, Nicolaides KH. Aspirin for the prevention of preterm and term preeclampsia: systematic review and metaanalysis. Am J Obstet Gynecol. 2018 Mar;218(3):287-293.e1. doi: 10.1016/j.ajog.2017.11.561. Epub 2017 Nov 11. PMID 29138036

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Started | 65 | 68 | 75
Completed | 57 | 54 | 68
Not Completed | 8 | 14 | 7
Not completed — Lost to Follow-up | 5 | 4 | 2
Not completed — Withdrawal by Subject | 3 | 6 | 3
Not completed — Discontinued Intervention | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg | Total
Number analyzed (Participants) | 65 | 68 | 75 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (6.3) | 29.6 (5.9) | 29.8 (6.1) | 29.7 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 68 | 75 | 208
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 9 | 26
  Not Hispanic or Latino | 57 | 59 | 66 | 182
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 2 | 2 | 5
  Black or African American | 6 | 9 | 14 | 29
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  White | 49 | 52 | 45 | 146
  More than one race | 0 | 2 | 3 | 5
  Hispanic | 8 | 3 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 65 | 68 | 75 | 208
BMI at enrollment [Mean (Standard Deviation); unit: kg/m2] | 29.2 (7.9) | 35.7 (10.0) | 34.1 (8.5) | 33.1 (9.2)
Method of Conception [Count of Participants; unit: Participants]
  Natural | 60 | 64 | 71 | 195
  Assisted by Ovulation Drugs | 3 | 3 | 2 | 8
  In Vitro Fertilization | 2 | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulsatility Index (PI)
Description: Uterine artery doppler is used to assess impedance to flow in the uterine artery three times: 11-16 weeks gestation(baseline), 18-22 weeks gestation (event 2), 28-32 weeks gestation (event 3). Data reported as change between 11-16 weeks gestation (baseline) and either 18-22 weeks gestation (event 2) or 28-32 weeks gestation (event 3).
  difference in uterine artery pulsatility index (PI) is calculated as the difference in PI for each patient between each trimester visit. PI at each visit will be calculated by averaging left-side and right-side PIs from each of three (or all available) images on each side for each patient using ultrasound technology. Unit of measure is a ratio: difference between the peak systolic and end-diastolic velocities divided by the mean flow velocity Relative change in uterine artery pulsatility index is a measure of flow to the uterus. A greater difference from the baseline value represents a greater improvement in placental perfusion.
Time Frame: Three times between 11 and 32 weeks of gestation.
Population: Participants delivered or lost to follow up not included
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 55 | 52 | 66
ratio
  Baseline to Event 2 | -0.56 (0.55) | -0.53 (0.34) | -0.43 (0.34)
  Baseline to Event 3: number analyzed (Participants) | 54 | 51 | 63
  Baseline to Event 3 | -0.88 (0.56) | -0.72 (0.41) | -0.58 (.54)

2. Secondary Outcome: Onset of Pre-eclampsia
Description: Frequency of Disease during pregnancy and postpartum as defined by American College of Obstetrics and Gynecology (ACOG) criteria
Time Frame: From enrollment at 11 weeks throughout pregnancy and postpartum ( 6 weeks after delivery), approximately 35 weeks
Population: Participants delivered or lost to follow up not included
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 58 | 61 | 73
Participants | 1 | 8 | 13

3. Secondary Outcome: Severity of Pre-eclampsia
Description: Frequency women are identified with Severe Features of the disease
Time Frame: From enrollment at 11 weeks throughout pregnancy and immediate postpartum ( 6 weeks after delivery), approximately 35 weeks
Population: Participants delivered or lost to follow up not included
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 58 | 62 | 73
Participants | 0 | 0 | 0

4. Secondary Outcome: Composite Neonatal Outcomes Including Frequency of Intraventricular Hemorrhage (IVH), Bronchopulmonary Dysplasia (BPD), Respiratory Distress Syndrome (RDS), Necrotising Enterocolitis(NEC)
Description: Frequency of adverse neonatal outcomes
Time Frame: Neonatal period ( first 28 days after birth)
Population: Participants lost to follow up not included
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 57 | 59 | 70
Participants | 5 | 17 | 21

5. Secondary Outcome: Change in s-ICAM Levels Over Time
Description: Serial biologic samples will be obtained in the first (baseline), second (event 2), and third (event 3) trimesters to measure changes in soluble Intercellular Adhesion Molecule (s-ICAM) levels over time.
Time Frame: Three times between 11 and 32 weeks of gestation
Population: Serum specimens were not collected for all patients at individual timepoints related to issues such as patient refusal for venipuncture. Some elected to discontinue participation
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 57 | 53 | 64
ng/ml
  Baseline and Event 2 | 6.1 (12.6) | 1.6 (30.8) | 7.9 (28.5)
  Baseline and Event 3: number analyzed (Participants) | 50 | 50 | 50
  Baseline and Event 3 | -29.6 (15.0) | -43.6 (32.2) | -34.1 (25.5)

6. Secondary Outcome: Change in PIGF Levels Over Time
Description: Serial biologic samples will be obtained in the first (baseline), second (event 2), and third (event 3) trimesters to measure changes in placental growth factor (PIGF) levels over time.
Time Frame: Three times between 11 and 32 weeks of gestation
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 57 | 53 | 64
pg/ml
  Baseline and Event 2 | 570.6 (377.8) | 568.3 (545.8) | 509.7 (457.8)
  Baseline and Event 3: number analyzed (Participants) | 51 | 50 | 50
  Baseline and Event 3 | -36.4 (69.3) | 1.0 (136.0) | -16.7 (44.1)

7. Secondary Outcome: Change in CRP Levels Over Time
Description: Serial biologic samples will be obtained in the first, second, and third trimesters to measure changes in C-reactive protein (CRP) levels over time.
Time Frame: Three times between 11 and 32 weeks of gestation
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 57 | 53 | 64
mg/L
  Baseline and Follow Up 1 | -0.5 (8.8) | 0.2 (9.3) | -2.7 (8.8)
  Baseline and Delivery: number analyzed (Participants) | 51 | 50 | 50
  Baseline and Delivery | -10.6 (11.9) | -13.4 (12.4) | -11.9 (13.2)

8. Secondary Outcome: Change in IL-6 Over Time
Description: Serial biologic samples will be obtained in the first, second, and third trimesters to measure changes in interleukin 6 (IL-6) levels over time.
Time Frame: Three times between 11 and 32 weeks of gestation
Population: Not enough serum from samples to run these measures
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change in TNF Over Time
Description: Serial biologic samples will be obtained in the first, second, and third trimesters to measure changes in tumor necrosis factor (TNFα) levels over time.
Time Frame: Three times between 11 and 32 weeks of gestation
Population: Not enough serum from samples to run these measures
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Gestational Age at Delivery
Description: measured in weeks, from the first day of the last menstrual cycle to delivery
Time Frame: At Delivery, up to 41 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
Number analyzed (Participants) | 65 | 68 | 75
weeks | 38.8 (1.3) | 36.0 (4.3) | 36.2 (4.7)

ADVERSE EVENTS:
Time Frame: 29 weeks
Description: Adverse Events were assessed from enrollment until delivery
Arm/Group | Control Group | Acetylsalicylic Acid 81mg | Acetylsalicylic Acid 162mg
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/68 | 0/75
Serious Adverse Events (participants affected / at risk) | 8/65 | 12/68 | 15/75
Other Adverse Events (participants affected / at risk) | 3/65 | 3/68 | 2/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=65) | Acetylsalicylic Acid 81mg (N=68) | Acetylsalicylic Acid 162mg (N=75)
Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 8 | 7 | 9
Intrauterine Fetal Demise (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 1
Placental Abruption (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 2
Previable Delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=65) | Acetylsalicylic Acid 81mg (N=68) | Acetylsalicylic Acid 162mg (N=75)
headaches (Nervous system disorders) | 2 | 0 | 0
Nose bleeds (Blood and lymphatic system disorders) | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0
Emesis (Gastrointestinal disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT03893630/Prot_SAP_000.pdf